CLINICAL TRIAL: NCT03288727
Title: Incidental Findings Produced by Diagnostic HTS: From the Needs of Patients to Organisational Considerations
Brief Title: Secondary Findings From High-throughput Sequencing: How to Announce Them With Respect to the Patient's Needs
Acronym: FIND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: OLIVIER-FAIVRE PREPS 2016
Record Dates: First submitted 2017-09-18; First posted 2017-09-20 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Development Disorders
MeSH Terms: interventions — Interviews as Topic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Negative IF result (Experimental)
  Interventions: Other: interviews with a psychologist
- Positive IF result (Experimental)
  Interventions: Other: interviews with a psychologist

INTERVENTIONS:
Other: interviews with a psychologist — an interview with a psychologist / sociologist will take place after completion of the on-site questionnaires to find out the reasons for their choice of accessing their secondary data and their experiences with the secondary data reported.

SUMMARY:
High-throughput whole-genome sequencing (WGS) is bringing new opportunities in the diagnosis of rare diseases. It will more frequently lead to a primary diagnosis (aim of the genetic consultation), but it may also lead to the discovery of mutations not related to the patient's disease. These findings are called "incidental findings" (IF) and may give rise to preventive or curative interventions in a personalised medicine approach.

The question of proposing to patients access to all or part of these findings is a matter of debate in France and elsewhere. This question has given rise to new challenges and new needs that professionals must respond to by implementing appropriate management and new skills. It raises specific ethical issues, which require precise understanding of the expectations and experiences of patients. Patients' diagnostic trajectories must also meet criteria for efficacy and financial and organisational sustainability for the healthcare establishments and, for the healthcare system. Our project aims to assess the expectations of patients/parents with regard to this opportunity, and to determine how information should be provided to patients and how they should be accompanied to ensure efficient and appropriate management.

ELIGIBILITY:
Inclusion Criteria:

* Adults or parents of of deceased foetuses/children (alive or deceased) or adults living under guardianship or deceased, with Development Disorders(DD) who will undergo WES for the first time for diagnostic purposes
* Consent to take part in the study
* Desire to screen for at least one group of IF
* Able to speak fluent French.

Exclusion Criteria:

* Patients withough national health insurance cover
* Absence of consent from the patient or his/her legal representative

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 342 (Actual)
Dates: Start 2017-11-13 (Actual); Primary Completion 2021-11-24 (Actual); Study Completion 2021-11-24 (Actual)

PRIMARY OUTCOMES:
Questionnaires on the expectations of patients/parents with regard to incidental findings (IF) | first day of the study
1) Questionnaires on their experience following the disclosure of IF (positive and negative), and their perception, needs and expectations with regard to the way the results are given. | at 6 months after the inclusion
2) Questionnaires on the repercussions of access to IF, in terms of experience/ appropriation of the results, needs and expectations in terms of accompaniment following disclosure of the results, and the recourse to care. | at 12 months after the inclusion

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - CHU Dijon Bourgogne, Dijon
  - Hospices Civils de Lyon, Lyon
  - Groupe Hospitalier Pitié-Salpêtrière, Paris